CLINICAL TRIAL: NCT05388305
Title: Clinical Study of Universal CAR-γδT Cell Injection in the Treatment of Refractory and Relapsed AML Patients
Brief Title: Universal CAR-γδT Cell Injection in the AML Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR-γδT for AML
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: AML

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR--γδT (Experimental)
  Interventions: Biological: CAR--γδT cells

INTERVENTIONS:
Biological: CAR--γδT cells — Biological: CAR-γδT; Drug:

SUMMARY:
To evaluate the safety of general-purpose CAR-γδT cells in patients with refractory post-transplant relapsed AML.

DETAILED DESCRIPTION:
To evaluate the efficacy and in vivo dynamics of general-purpose CAR-γδT cells in the treatment of refractory relapsed AML patients, and to explore the appropriate therapeutic dose and delivery mode.

ELIGIBILITY:
Inclusion Criteria:

* The clinical diagnosis was difficult to treat recurrent acute myeloid leukemia；
* Flow cytometry (FCM) or immunohistochemistry of tumor~ cells confirmed positive expression of CD123；
* 18 years old ≤ age ≤70 years old;
* The expected survival from the date of informed consent is more than 3 months;
* ECOG≤2;
* The functions of vital organs shall meet the following conditions:

  1) EF>50%, and no obvious ECG abnormality; 2) SpO2 90% or more; 3) Cr 2.5 ULN or less; 4) ALT And AST≤5ULN, TBil≤3ULN;
* Subjects who plan to become pregnant must agree before study enrollment and after study duration of 6 months Use contraception; Inform the investigator immediately if the subject is pregnant or suspected to be pregnant;
* Subject or guardian understands and signs the informed consent.

Exclusion Criteria:

* Other diseases that have not been effectively controlled, including but not limited to persistent or poorly controlled infections and diseases Congestive heart failure, unstable angina pectoris, arrhythmias, poorly controlled lung disease Or mental illness;
* Other active malignant tumors;
* Complicated with severe infection that cannot be effectively controlled;
* Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive, peripheral blood hepatitis B virus (HBV)DNA higher than the detection limit should be excluded; If hepatitis C virus (HCV) antibody positive, peripheral blood HCV RNA positive need to be eliminated; Cytomegalovirus (CMV)DNA positive; Epstein-barr virus DNA in peripheral blood was positive;
* Human immunodeficiency virus (HIV) infection or syphilis infection;
* Have a history of severe allergy to biological products (including antibiotics);
* Acute graft-versus-host reaction (GVHD) was still present one month after discontinuation of immunosuppressant therapy Allogeneic hematopoietic stem cell transplantation patients;
* Female subjects are in pregnancy and lactation;
* Active autoimmune diseases requiring systemic immunosuppression;
* Conditions that the investigator believes may increase the risk of the subject or interfere with the results of the test;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence and severity of adverse events | First 1 month post CAR-T cells infusion
  To evaluate the possible adverse events occurred within first one month after CAR-γδT infusion, including the incidence and severity of symptoms such as cytokine release syndrome and neurotoxicity

CONTACTS AND LOCATIONS:
Overall Officials: Liang Huang, PhD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No